CLINICAL TRIAL: NCT01036529
Title: Spinal Cord Stimulation With Precision® Spinal Cord Stimulation System Versus Reoperation for Failed Back Surgery Syndrome
Brief Title: Spinal Cord Stimulation With Precision® System Versus Reoperation for Failed Back Surgery Syndrome
Acronym: Evidence
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Closed due to continued slow enrollment.
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A2005
Record Dates: First submitted 2009-12-17; First posted 2009-12-21 (Estimated); Results first posted 2013-10-28 (Estimated); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Failed Back Surgery Syndrome; Pain; Back Pain
Keywords: Spinal Cord Stimulation; Decompression; Fusion with or without instrumentation; Discectomy; Laminectomy; Laminotomy; Foraminotomy
MeSH Terms: conditions — Failed Back Surgery Syndrome; Pain; Back Pain | interventions — Diskectomy; Laminectomy; Foraminotomy; Gene Fusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Precision Spinal Cord Stimulator (Experimental): Spinal Cord Stimulation
  Interventions: Device: Precision Spinal Cord Stimulator
- Back Surgery (Active Comparator): Discectomy, laminotomy, laminectomy, foraminotomy, fusion with or without instrumentation
  Interventions: Procedure: Back Surgery

INTERVENTIONS:
Device: Precision Spinal Cord Stimulator — Programming settings will be specific to the individual needs in accordance with the labeling
  Arms: Precision Spinal Cord Stimulator
Procedure: Back Surgery — Different types of back surgery may be performed
  Other Names: Discectomy; Laminotomy; Laminectomy; Foraminotomy; Foraminectomy; Fusion with or without instrumentation
  Arms: Back Surgery

SUMMARY:
The EVIDENCE trial is a randomized controlled trial comparing the therapeutic effectiveness and cost-effectiveness of the Precision® Spinal Cord Stimulation with that of reoperation as a treatment of pain in patients with Failed Back Surgery Syndrome (FBSS). FBSS is defined as persistent or recurrent pain following one or more lumbosacral spine surgical procedures. Surgical procedures that can result in FBSS can be categorized as either decompression or decompression followed by fusion with or without instrumentation. The pain of FBSS is categorized as neuropathic, which involves pathological nerve activity and is commonly characterized by patients as shooting or burning and/or nociceptive, which signals actual or impending tissue damage or inflammation.

DETAILED DESCRIPTION:
The co-primary study endpoints are proportion of subjects with ≥50% leg pain relief without crossover at 6 and at 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Primary pain type - neuropathic with concordant radicular or neurological findings
* Significant complaint of persistent or recurrent radicular leg pain, with or without low back pain
* One or more prior lumbosacral surgical procedures (no upper limit)
* At least 6 months duration of persistent or recurrent radicular leg pain, with or without low back pain
* Study candidates meet the criteria for a specific surgical intervention as recorded by a surgeon: pain refractory to conservative care, with concordant neurologic, tension, and/or mechanical signs and imaging findings of surgically remediable neural compression
* MRI or CT myelogram of the lumbar and thoracic spine (within 12 months prior to screening) that rules out pathology that might compromise SCS electrode placement or pathology, in addition to neural compression, that might contribute to the subject's pain
* All study candidates must pass study site's routine psychological/psychiatric evaluation for SCS before randomization to SCS or reoperation
* At least 18 years of age
* Subject signs informed consent

Exclusion Criteria:

* Chief complaint of mechanical low back pain (e.g. pain that a recumbent position relieves completely)
* Pain intensity of always 10 on a 0-10 Numerical Rating Scale over the past 6 months based on subject recall
* Radiographic evidence of frank instability (grossly mobile spondylolisthesis or abnormal subluxation) requiring fusion, calcific arachnoiditis, or severe thoracic stenosis
* Radiographically demonstrated (by myelographic block or its MRI equivalent) critical cauda equinal compression
* A disabling or potentially disabling neurologic deficit (e.g., foot drop, neurogenic bladder) in the distribution of a nerve root or roots caused by surgically remediable compression
* A predominance of non-organic signs on physical exam
* A concurrent clinically significant or disabling chronic pain problem or condition that is likely to confound evaluation of study endpoints (e.g., chronic migraine, significant arthrosis of the hip associated with groin pain as primary complaint)
* Significant substance abuse issues
* Major untreated psychiatric comorbidity
* Unresolved issues of secondary gain (e.g., litigation)
* Expected inability to report treatment outcome adequately
* Expected inability to operate SCS system
* Pregnancy (actual or planned)
* Life expectancy less than 3 years due to other serious medical condition(s)
* Active local or systemic infection
* Prior SCS procedure
* Presence of intrathecal drug pump
* Participation in another clinical study that would confound data of this study
* Occupational risk that would rule out SCS
* Medical or cardiac condition(s) or therapies, or foreseeable need for therapies or diagnostic tests (e.g., MRI), that preclude SCS and/or reoperation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard North, M.D., Principal Investigator — The Sandra and Malcolm Berman Brain & Spine Institute
Locations (18):
- United States (13):
  - Scripps Clinic, La Jolla, California
  - University of California San Diego, La Jolla, California
  - Orthopedic Research Foundation, Savannah, Georgia
  - Millenium Pain Center, Bloomington, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - The University of Illinois Medical Center, Chicago, Illinois
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - St. Patrick Hospital, Missoula, Montana
  - The Center for Clinical Research, LLC, Winston-Salem, North Carolina
  - Geisinger Medical Center, Danville, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Swedish Neuroscience Institute, Seattle, Washington
  - Pacific Medical Center, Seattle, Washington
- Canada (2):
  - Hopital de Enfant-Jesus, Québec, Quebec
  - Regina General Hospital, Regina, Saskatchewan
- CHU de Nantes-Hopital Laennec, Nantes, France
- United Kingdom (2):
  - Frenchay Hospital, Bristol
  - James Cook University Hospital, Middlesbrough

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited for participation from February 2010 to June 2012.
Pre-assignment Details: A total of 274 subjects were screened for participation.After screening, 75 subjects were eligible for participation. Of the eligible subjects, 47 declined randomization. A total of 28 subjects were randomized.
Groups:
- Precision Spinal Cord Stimulator: Precision Spinal Cord Stimulator Intervention
Period: Overall Study
Arm/Group | Precision Spinal Cord Stimulator | Back Surgery
Started | 13 | 15
Baseline Visit | 10 | 13
Index Procedure | 10 (Index Procedure: Trial Stimulation) | 11 (Index Procedure: Surgery)
3 Month Follow-up | 7 | 9
6 Month Follow-up | 6 | 7
12 Month Follow-up | 4 | 3
Requested Crossover | 1 | 2
Crossover to Other Group | 1 | 1
Completed | 0 | 0
Not Completed | 13 | 15
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Sponsor study termination | 11 | 12

BASELINE CHARACTERISTICS:
Population: This represents the number of subjects with demographic information provided at enrollment (collected before baseline visit).
Groups:
- Precision Spinal Cord Stimulator: Precision Spinal Cord Stimulation System
- Total: Total of all reporting groups
Arm/Group | Precision Spinal Cord Stimulator | Back Surgery | Total
Number analyzed (Participants) | 11 | 14 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (12) | 57 (15.3) | 54.9 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 4 | 10 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 7 | 12 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Showing ≥50% Self-reported Leg Pain Relief From Baseline Without Request for Crossover to the Other Treatment
Time Frame: 3, 6- and 12- months post-index procedure
Measure: Number; unit: proportion of participants
Arm/Group | Precision Spinal Cord Stimulator | Back Surgery
Number analyzed (Participants) | 7 | 9
proportion of participants
  3 Month (7 subject Stimulation, 9 Subjects Surger) | 0.86 | 0.44
  6 Month (6 subjects for Stimulation and Surgery) | 0.5 | 0.5
  12 month (4 subjects for Stim, 3 subjects Surgery) | 1.0 | 0.33

ADVERSE EVENTS:
Description: The adverse events for all subjects (including cross-over subjects) were collected within the group that each subject was originally randomized.
Arm/Group | Precision Spinal Cord Stimulator | Back Surgery
Serious Adverse Events (participants affected / at risk) | 1/13 | 4/15
Other Adverse Events (participants affected / at risk) | 3/13 | 2/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Precision Spinal Cord Stimulator (N=13) | Back Surgery (N=15)
Radicular Pain (Nervous system disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Sternal Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Precision Spinal Cord Stimulator (N=13) | Back Surgery (N=15)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 1 (1)
Implant site haematoma (General disorders) | 1 (1) | 0 (0)
Implant site pain (General disorders) | 1 (1) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site pruritis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated early due to slow enrollment. Only 28 of the 200 planned subjects were enrolled. Based on the small numbers and early termination, the primary outcome measures were not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No